CLINICAL TRIAL: NCT05454358
Title: Letrozole as Maintenance Therapy Versus Observation After Adjuvant Treatment on the Prognosis for Post-surgical Endometrial Cancer Patients With Non-specific Molecular Profile: a Superiority Randomized Controlled Trial
Brief Title: Letrozole as Maintenance Therapy for Post-surgical Endometrial Cancer Patients With NSMP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: No enough participants
Sponsor: Fudan University (Other)
Collaborators: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Xiaojun Chen, Vice President of Obstetrics and Gynecology Hospital of Fudan University, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-54
Record Dates: First submitted 2022-06-26; First posted 2022-07-12 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; letrozole; maintenance therapy; molecular classification; non-specific molecular profile
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole (Experimental): Letrozole 0.5mg qd po for 2 years after postoperative adjuvant therapy
  Interventions: Drug: Letrozole 2.5mg
- Observation (No Intervention): Observation alone without any other therapy after postoperative adjuvant therapy

INTERVENTIONS:
Drug: Letrozole 2.5mg — Letrozole 0.5mg qd po for 2 years after postoperative adjuvant therapy
  Other Names: Letrozole 2.5mg qd po for 2 years
  Arms: Letrozole

SUMMARY:
Aim to investigate the effect of Letrozole as maintenance after adjuvant treatment on the prognosis of post-operative endometrial cancer patients with non-specific molecular profile.

DETAILED DESCRIPTION:
This is an open label multi-center superiority randomized controlled trial, aimed to investigate the effect of Letrozole as maintenance therapy on the prognosis of post-operative endometrial cancer patients with non-specific molecular profile.

The molecular classification of non-specific molecular profile (NSMP) is the most common type of endometrial cancer. Reducing the recurrence rate and improving the survival rate in patients with NSMP can effectively improve the overall prognosis of endometrial cancer.

NSMP endometrial cancers are featured as high sensitivity to hormones, which could be a potential target to improve the prognosis. Antiestrogenic therapy might be an effective treatment to improve the prognosis of NSMP endometrial cancer with high risk of recurrence and metastasis.

Letrozole, an oral non-steroidal aromatase inhibitor, might have positive impact on those patients as maintenance therapy after first-line postoperative adjuvant treatments. The current standardized treatment for intermediate-high risk endometrial cancer patients after chemotherapy and radiotherapy includes none but observation alone. However, with little adverse effects, low cost and easy availability, the practice of letrozole in hormonally-responsive breast cancer after surgery added to evidence to have an improvement in the prognosis in intermediate-high risk endometrial cancer. Thus, it is necessary to carry out a randomized trial to investigate the role of letrozole as maintenance therapy after postoperative adjuvant treatment in the prognosis of intermediate-high risk endometrial cancer.

This study were approved by the Ethics Committees of Obstetrics and Gynecology Hospital of Fudan University and all other institutes. Before initiation of study procedures, written informed consent will be obtained from each patient regarding risks of treatments and agreement of using their clinical data for research purpose.

This is a multicentered, open-label, randomized clinical trial. Randomization will be carried out in each center. A computer-based procedure of simple randomization (SPSS for Mac, version 22.0; IBM ) will be used for participant enrollment and randomization. Before an individual is successfully enrolled, her treatment assignment will remain concealed. This trial will be open label: patients and study physicians were aware of treatment assignment.

Patients will be stratified into 3 groups by operative staging (FIGO 2009), pre- and post- operative imaging assessment and residual tumor condition after surgery: stage I/II without early postoperative residues, stage III/IV without late postoperative residues and patients with postoperative residues. Eligible patients in each stratification of each center will be randomly assigned (1:1) to receive:

Arm 1. Letrozole 0.5mg qd po for 2 years after postoperative adjuvant therapy, or Arm 2. Observation alone without any other therapy after postoperative adjuvant therapy.

A definitive surgery should be performed after the latest NCCN guidelines, including a hysterectomy with/without bilateral salpingo-oophorectomy plus sentinel node biopsy or pelvic lymph node sampling with para-aortic lymph node sampling.

All the patients must meet the criteria to have postoperative adjuvant treatments, excluding patients with low prognostic risk: stage IA endometrioid + low-grade* +lymphovascular space invasion (LVSI) negative or focal, or those requiring no adjuvant therapy after surgery. Postoperative adjuvant treatments are carried out following the latest NCCN or ESGO guidelines according to doctors' choice.

Molecular classification must be performed and proved be to non-specific molecular profile (NSMP) according to diagnostic algorithm for the integrated histomolecular endometrial carcinoma classification (WHO classification of tumors, 5th edition, female genital tumours).

Statistical analyses On the basis of data from previous studies (Molecular Classification of PORTEC-3 Trial；GOG-249；GOG-99), the 3-year PFS is expected to be 80% in the observation group. Letrozole as maintenance therapy would improve 3-year PFS to 90%, which is considered as superior to observation alone. An accrual of 299 patients in 3 years will provide the study with adequate power (90%) to detect a clinically relevant absolute difference of 10% in 3-year PFS (90% vs 80%) between both groups (one-sided test, a=0.05), with a lost follow up rate ≤10%. Analyses will be done firstly by intention to treat.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 18 years old;
2. Initial diagnosed with stage I-IV(FIGO2009) endometrial epithelial cancer, regardless of pathological types;
3. Surgery must have included a hysterectomy, bilateral salpingo-oophorectomy and sentinel node biopsy; pelvic lymph node sampling and para-aortic lymph node sampling are optional;
4. Life expectancy of 2 or more years.
5. Confirmed NSMP with intermediate or higher prognostic risk according to post-operative clinical pathological assessment and molecular classification;

   1. Intermediate prognostic risk group:

      * Stage lB endometrioid + Iow-grade* + LVSI negative or focal
      * Stage IA endometrioid + high-grade*+ LVSI negative or focal
      * Stage IA non-endometrioid (serous, clear cell, undifferentiated carcinoma, carcinosarcoma, mixed) without myometrial invasion
   2. High-intermediate prognostic risk group:

      * Stage I endometrioid + substantial LVSI, regardless of grade and depth of invasion
      * Stage lB endometrioid high-grade*, regardless of LVSI status
      * Stage II
   3. High prognostic risk group:

      * Stage Ill-IVA with no residual disease
      * Stage I-IVA non-endometrioid (serous, clear cell, undifferentiated carcinoma, carcinosarcoma, mixed) with myometrial invasion, and with no residual disease
   4. Advanced Metastatic:

      * Stage III-IVA with residual disease
      * Stage IVB Low grade: G1-2; High grade:G3;
6. Received conventional adjuvant therapy after surgery according to the latest version of NCCN or ESGO/ESTRO/ESP guidelines;
7. Patients with residual tumor after surgery (any single site) must have achieved complete response or partial response after post-operative adjuvant therapy;
8. Expected start of letrozole maintenance within 3 months after adjuvant therapy;
9. Adequate organ function as defined by the following criteria:

   * White blood cell (WBC) ≥ 3000/μL or Absolute neutrophil count (ANC) ≥1500/μL
   * Platelets ≥100,000/μL
   * Serum Aspartate transaminase (AST) and/or serum alanine transaminase (ALT) ≤ 2 times upper limit of normal (ULN)
   * Serum creatinine ≤2 times ULN
10. Karnofsky score ≥60;
11. Eastern Cooperative Oncology Group (ECOG) Performance status ≤2;
12. Ability to take anti-thyroid drugs, calcium, vitamin D or bisphosphonates together.

Exclusion Criteria:

1. Endometrial stromal tumor;
2. Recurrent endometrial cancers;
3. Patients with low prognostic risk according to post-operative clinical pathological assessment ( Stage IA endometrioid + low-grade* +LVSI negative or focal);
4. Patients require no adjuvant therapy after surgery;
5. Negative expression in estrogen receptor or progesterone receptor according to post-operative Immunohistochemistry;
6. Received other adjuvant therapy within 6 months before surgery: including neoadjuvant therapy, hormone therapy, targeted therapy, immunotherapy and biotherapy, etc;
7. Patients with contraindications for letrozole;
8. Patients with other malignant tumors;
9. History of vital organ transplantation;
10. History of immune disease and need to take immunosuppressor;
11. Uncontrolled psychiatric illness or other situations that would limit compliance with study requirements;
12. History of drug abuse;
13. Participated in other clinical trials;
14. No ability or intention to receive letrozole maintenance/sign the consent/obey the study requirements.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
the 3-year Progression-Free-Survival(PFS) | 3 years
  The percentage of patients who have first relapse within 3 years after surgery

SECONDARY OUTCOMES:
the 3-year Overall survival(OS) | 3 years
  The percentage of patients who died within 3 years after surgery.
the 5-year PFS and OS | 5 years
  The percentage of patients who have first relapse within 5 years after surgery. The percentage of patients who died within 5 years after surgery.
Incidence of adverse events | From date of recruitment, assessed up to 5 years
  Adverse events related with intervention. Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 will be recorded, as well as incidence of adverse events.
Quality of life change | baseline, 1 year, and 2 years
  Collect the questionnaire EORTC QLQ-C30 V3.0-EN24 and questionnaire MENQOL, and count scores change through intervention (Letrozole or Observation).
Site of recurrence | 8 years
  The frequency of recurrence site in different groups.

OTHER OUTCOMES:
Recurrence related factors | 8 years
  Recurrence related clinical pathological factors and molecular biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojun Chen, Ph.D, M.D, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, China